CLINICAL TRIAL: NCT00346931
Title: Phacotrabeculotomy vs. CCI+Phaco in Patients With Borderline Control of Intraocular Pressure
Brief Title: Phacotrabeculotomy Versus CCI+Phaco in Patients With Borderline Control of Intraocular Pressure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof. Dr. Clemens Vass, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCI-PTO-2004-AKH
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2006-06

CONDITIONS: Primary Open Angle Glaucoma; Pseudoexfoliative Glaucoma
Keywords: glaucoma; cataract; surgery; intraocular pressure; phacoemulsification; trabeculotomy
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Cataract | interventions — Phacoemulsification; Lens Implantation, Intraocular; Trabeculectomy

INTERVENTIONS:
Procedure: Phacoemulsification, implantation of intraocular lens
Procedure: Phacoemulsification, Implantation of IOL, trabeculotomy

SUMMARY:
The purpose of the study is to determine whether combined cataract and glaucoma surgery (phacotrabeculotomy)is more effective in lowering intraocular pressure than cataract surgery alone in patients with borderline control of intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Primary Open Angle or Pseudoexfoliative Glaucoma and Cataract

Exclusion Criteria:

* Other glaucoma than POAG or PEX-Glaucoma
* Medically uncontrolled Glaucoma:

IOP > 24 mmHg with two topical medications IOP > 21 mmHg with three topical medications

* IOP < 18 mmHg with two topical medications IOP < 16 mmHg with three topical medications
* previous ocular surgery
* other ocular pathologies affecting visual acuity
* disorders of immune system

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Constant Intraocular Pressure <18 mmHg with/without medication

SECONDARY OUTCOMES:
Number of Patients with Constant Intraocular Pressure <18 mmHg without medication
Number of Patients with Constant Intraocular Pressure <21 mmHg with/without medication
Number of Patients needing surgical retreatment
Number of Patients with failure of surgical retreatment
Mean IOP after 1 and 2 years
Mean number of medication after 1 and 2 years
Number of intraoperative complications
comparison of postoperative complications between the groups
Visual acuity
decrease in perimetry

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Vass, Univ.Prof.Dr.med.univ., Principal Investigator — Medical University of Vienna